CLINICAL TRIAL: NCT05856266
Title: An 18-month Low-interventional Prospective, Multicentre Study to Assess Joint Outcomes in Patients With Haemophilia A or B on Prophylaxis With Efmoroctocog Alfa or Eftrenonacog Alfa
Brief Title: An 18-month Low-interventional Study to Assess Joint Health in Haemophilia A and B Patients on Prophylaxis With Efmoroctocog Alfa or Eftrenonacog Alfa
Acronym: JOIN-us
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The Sponsor has decided to stop the phase 4 study Sobi.HAEM89-007 (JOIN-us) due to a realignment of its development activities.
  The clinical trial hasn't been terminated due to a change in the benefit-risk balance.
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: IQVIA Pvt. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Sobi.HAEM89-007; 2022-502921-16-00 (Other: EU Drug Regulatory Authorities Clinical Trial System)
Record Dates: First submitted 2023-04-24; First posted 2023-05-12 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: Blood coagulation disorder; Coagulation protein disorder; Haemophilia; FVIII; FIX; Efmoroctocog alfa; Eftrenonacog alfa
MeSH Terms: conditions — Hemophilia A; Hemophilia B; Blood Coagulation Disorders; Coagulation Protein Disorders | interventions — High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: This is a low-interventional study, with the drugs being prescribed and used according to clinical practice.
  The interventions in the study are the addition of the mandatory joint examinations HEAD-US (ultrasound) and HJHS (functional joint assessment).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Efmoroctocog alfa or eftrenonacog alfa (Other): Efmoroctocog alfa or eftrenonacog alfa is prescribed and used according to usual clinical practice.
  Interventions: Procedure: Haemophilia Early Arthropathy Detection with Ultrasound (HEAD-US); Other: Haemophilia Joint Health Score (HJHS)

INTERVENTIONS:
Procedure: Haemophilia Early Arthropathy Detection with Ultrasound (HEAD-US) — Ultrasound examination
Other: Haemophilia Joint Health Score (HJHS) — Functional joint examination

SUMMARY:
The goal of this low-interventional study is to describe the overall joint health in patients with haemophilia A or haemophilia B prophylactically treated with rFVIIIFc or rFIXFc.

The main question it aims to answer is the:

• Evaluation of the overall joint status as detected by ultrasound in haemophilia A and B patients treated with rFVIIIFc or rFIXFc prophylaxis over the 18-month study period.

Participants will come to 6-monthly visits during the 18-month long study period and will perform an ultrasound with the Haemophilia Early Arthropathy Detection with Ultrasound (HEAD-US) protocol at each visit. At baseline and end of study visits, the patients will be assessed with the clinical scoring system Haemophilia Joint Health Score (HJHS) and complete patient questionnaires. Retrospective data from patient medical records will also be collected for at least 6 months before enrolment in the study.

DETAILED DESCRIPTION:
The main purpose of this study is to prospectively describe the joint health over an 18-month period of prophylactic treatment with rFVIIIFc or rFIXFc in patients with haemophilia A or haemophilia B in a real-world setting in Europe.

This is a low-interventional, multicentre study using point-of-care US examination for regular monitoring of joint health and detection of hypertrophic synovium, cartilage and bone damage. At the same time, clinical joint status will also be examined by HJHS. This study will evaluate the presence, resolution, recurrence, and new development of target joints. It will also describe bleeding episodes and evaluate the quality of life and physical activity with PROs. If patients are using the CE marked Florio HAEMO app in their routine clinical practice, they will be offered to participate in an optional sub-study that aims to explore possible correlations between the levels of physical activity, the estimated FVIII/FIX levels and bleeding occurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 6 years
2. Diagnosis of haemophilia A or B
3. Having at least 6 months documented pre-study treatment data regarding treatment prescriptions and bleeding episodes prior to the baseline visit
4. Previous treatment for haemophilia A or B with any marketed recombinant and/or plasma-derived FVIII or FIX concentrate for at least 6 months
5. Start of prophylactic treatment with rFVIIIFc or rFIXFc prior to study enrollment or latest at the baseline visit, in accordance with local regulations
6. Signed and dated informed consent provided by the patient, or the patient's legally authorized representative for patients under the legal age. Assent should be obtained from paediatric patients in accordance with local regulations

Exclusion Criteria:

1. Any medical condition which in the opinion of the investigator makes the subject patient unsuitable for inclusion
2. Prophylactic treatment with non-factor therapy during the 6 months prior to enrolment
3. Presence of factor VIII or FIX inhibitory antibodies (inhibitors) (≥0.60 Bethesda Units [BU]/mL) at the latest available inhibitor test
4. Enrolment in a concurrent clinical interventional study, or intake of an IMP, within three months prior to inclusion in this study
5. Foreseeable inability to cooperate with given instructions or study procedures

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Lethagen, MD, PhD, Study Director — Swedish Orphan Biovitrum AB (publ)
Locations (56):
- Bulgaria (2):
  - Study site 100, Sofia
  - Study site 101, Sofia
- Croatia (2):
  - Study site 102, Zagreb
  - Study site 103, Zagreb
- Czechia (5):
  - Study site 108, Brno
  - Study site 107, Liberec
  - Study site 104, Olomouc
  - Study site 105, Prague
  - Study site 106, Prague
- France (20):
  - Study site 115, Bordeaux
  - Study site 129, Caen
  - Study site 125, Chambéry
  - Study site 110, Clermont-Ferrand
  - Study site 123, Dijon
  - Study site 124, Lille
  - Study site 111, Lyon
  - Study site 126, Marseille
  - Study site 120, Nancy
  - Study site 121, Nantes
  - Study site 113, Nîmes
  - Study site 119, Paris
  - Study site 130, Paris
  - Study site 118, Poitiers
  - Study site 117, Reims
  - Sudy site 122, Rennes
  - Study site 109, Rouen
  - Study site 112, Strasbourg
  - Study site 128, Toulouse
  - Study site 114, Tours
- Study site 131, Budapest, Hungary
- Ireland (2):
  - Study site 132, Dublin
  - Study site 133, Dublin
- Italy (7):
  - Study site 136, Bologna
  - Study site 134, Brescia
  - Study site 138, Catania
  - Study site 140, Milan
  - Study site 137, Palermo
  - Study site 135, Pisa
  - Study site 139, Vicenza
- Romania (5):
  - Study site 145, Baia Mare
  - Study site 141, Bucharest
  - Study site 143, Craiova
  - Study site 146, Iași
  - Study site 142, Timișoara
- Study site 147, Ljubljana, Slovenia
- Spain (10):
  - Study site 151, A Coruña
  - Study site 150, Alicante
  - Study site 152, Barcelona
  - Study site 149, Madrid
  - Study site 154, Málaga
  - Study site 156, Oviedo
  - Study site 153, Salamanca
  - Study site 157, Valencia
  - Study site 155, Valladolid
  - Study site 158, Zaragoza
- Study site 159, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Efmoroctocog Alfa or Eftrenonacog Alfa
Started | 10
Completed (Study was terminated.) | 0
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Efmoroctocog Alfa or Eftrenonacog Alfa
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Romania | 1
  Czechia | 4
  France | 2
  Spain | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total HEAD-US Score up to Month 18 (End of Study - EOS)
Description: HEAD-US is a standardized, fast, repeatable, and simple ultrasound scoring protocol for hemophiliac joints.
  The HEAD-US joint score will be calculated for the six index joints (elbows, knees, and ankles). The specific joint score is made up of three item scores: disease activity (synovitis), disease damage of articular surfaces, and disease damage of subchondral bone. The specific joint score is the sum of the three item scores for each specific joint. Its values range from 0 (minimum) to 8 (maximum). The total score represents the sum of item scores for abnormalities detected.
Time Frame: Baseline and month 18
Population: No patient had any post baseline assessmen t
Arm/Group | Efmoroctocog Alfa or Eftrenonacog Alfa
Number analyzed (Participants) | 0

2. Secondary Outcome: Change From Baseline in HEAD-US Score for Hypertrophic Synovium
Description: HEAD-US is a standardized, fast, repeatable, and simple ultrasound scoring protocol for hemophiliac joints.
  The HEAD-US joint score will be calculated for the six index joints (elbows, knees, and ankles). The disease activity (synovitis) score rates the status of the hypertrophic synovium. Hypertrophic synovium is graded in three steps (0: absent/minimal; 1: mild/moderate [score=1], 2: severe [score=2]) based on the comprehensive evaluation of the joint recesses and the mean amount of synovial tissue contained in them.
Time Frame: Baseline, month 6, 12 and 18
Reporting Status: Not Posted

3. Secondary Outcome: Change From Baseline in HEAD-US Score for Cartilage
Description: HEAD-US is a standardized, fast, repeatable, and simple ultrasound scoring protocol for hemophiliac joints.
  The HEAD-US joint score will be calculated for the six index joints (elbows, knees, and ankles). Concerning the articular cartilage, the damage is graded in five steps (0: normal; 1: echotexture abnormalities and focal loss involving <25% of the target surface [score=1]; 2: partial/full-thickness loss of the cartilage involving at least 50% of the target surface [score=2]; 3: partial/full-thickness loss of the cartilage involving >50% of the target surface [score=3]; 4: complete cartilage destruction or absent visualization of the articular cartilage on the target surface [score=4]).
Time Frame: Baseline, month 6, 12 and 18
Reporting Status: Not Posted

4. Secondary Outcome: Change From Baseline in HEAD-US Score for Bone
Description: HEAD-US is a standardized, fast, repeatable, and simple ultrasound scoring protocol for hemophiliac joints.
  The HEAD-US joint score will be calculated for the six index joints (elbows, knees, and ankles). Damage of subchondral bone is scored using a three-grade scale (0: normal; 1: mild irregularities of the subchondral bone with/without initial osteophytes around the joint [score=1]; 2: deranged subchondral bone with/without erosions and presence of prominent osteophytes around the joint [score=2]).
Time Frame: Baseline, month 6, 12 and 18
Reporting Status: Not Posted

5. Secondary Outcome: Change From Baseline in Total Hemophilia Joint Health Score (HJHS) at Month 18 (EOS)
Description: The HJHS measures joint health, in the domain of body structure and function (i.e., impairment). The six index joints (elbows, knees, and ankles) will be examined and scored. The minimum score per joint is 0, the maximum score is 20. In addition, Gait is scored on a scale from 0 to 4 based on the number of skills that are not within the normal limits.
  The total score will be the sum of scores across all six joints plus the gait score (range from 0 to 124, with 0 being normal and 124 being the most severe disease).
Time Frame: Baseline and month 18
Reporting Status: Not Posted

6. Secondary Outcome: Number of Target Joints
Description: A target joint is defined as a joint with three or more spontaneous bleeds into the joint within a consecutive 6-month period. The study will evaluate the presence, resolution, recurrence, and new development of target joints.
Time Frame: Baseline, month 6, 12 and 18
Reporting Status: Not Posted

7. Secondary Outcome: Location of Target Joints
Description: as for outcome 6
Time Frame: Baseline, month 6, 12 and 18
Reporting Status: Not Posted

8. Secondary Outcome: Total Annualized Bleeding Rate (ABR)
Description: For any bleeding episode, the following will be collected: bleeding episode circumstance (e.g., spontaneous, traumatic), bleeding episode location (e.g., muscle, joint, other), date of bleeding episode, dose (IU) and number of injections used to treat the bleed.
Time Frame: 6 months retrospective period to baseline, baseline to 6 months, 6-12 months, 12-18 months and entire study period
Reporting Status: Not Posted

9. Secondary Outcome: Joint ABR
Description: For any bleeding episode, the following will be collected: bleeding episode circumstance (e.g., spontaneous, traumatic), bleeding episode location, date of bleeding episode, dose (IU) and number of injections used to treat the bleed.
Time Frame: 6 months retrospective period to baseline, baseline to 6 months, 6-12 months, 12-18 months and entire study period
Reporting Status: Not Posted

10. Secondary Outcome: Target Joint ABR
Description: as for outcome 9
Time Frame: 6 months retrospective period to baseline, baseline to 6 months, 6-12 months, 12-18 months and entire study period
Reporting Status: Not Posted

11. Secondary Outcome: Traumatic/Spontaneous ABR
Description: as for outcome 8
Time Frame: 6 months retrospective period to baseline, baseline to 6 months, 6-12 months, 12-18 months and entire study period
Reporting Status: Not Posted

12. Secondary Outcome: PROMIS Physical Function/Activity Short Form 6b and 8a Scores
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) is a validated system of reliable and precise measures of patient-reported health status. PROMIS measures cover physical, mental, and social health, use a 5-point Likert response scale and a recall period of the past 7 days. The Numeric Rating Scale measures for adults (6b) consist of a single item rating physical function on average over the past 7 days, ranging from 5 (without any difficulty) to 1 (unable to do). Lower scores mean a worse outcome.
  The Numeric Rating Scale measures for pediatric and parent proxy (8a) each consist of a single item rating physical activity on average over the past 7 days, ranging from 1 (no days) to 5 (6-7 days). Lower scores mean a worse outcome.
Time Frame: Baseline and 18 months
Reporting Status: Not Posted

13. Secondary Outcome: PROMIS Pain Intensity 3a and 1a Scores
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) is a validated system of reliable and precise measures of patient-reported health status. PROMIS measures cover physical, mental, and social health, use a 5-point Likert response scale and a recall period of the past 7 days. The Numeric Rating Scale measures for adults (3a) consist of a single item rating pain over the past 7 days from 1 (had no pain) to 5 (very severe). Higher scores mean a worse outcome. The Numeric Rating Scale measures for pediatric and parent proxy (1a) each consist of a single item rating pain over the past 7 days, ranging from 0 (no pain) to 10 (worst pain you can think of). Higher scores mean a worse outcome.
Time Frame: Baseline and month 18
Reporting Status: Not Posted

14. Secondary Outcome: PROMIS Pain Interference Short Form 6a and 8a Scores
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) is a validated system of reliable and precise measures of patient-reported health status. PROMIS measures cover physical, mental, and social health, use a 5-point Likert response scale and a recall period of the past 7 days. The Numeric Rating Scale measures (adult, pediatric, parent proxy) each consist of a single item rating pain interference with different activities over the past 7 days, ranging from 1 (not at all/never) to 5 (very much/almost always). Higher scores mean a worse outcome.
Time Frame: Baseline and month 18
Reporting Status: Not Posted

15. Secondary Outcome: IPAQ-SF Scores
Description: International Physical Activity Questionnaire - Short Form (IPAQ-SF). The IPAQ-SF is a validated, 7-day recall questionnaire measuring current levels of physical activity. Scoring of the IPAQ results in a continuous variable in the form of total MET-minutes per week, as well as categorization into high, moderate, or low physical activity level. Higher scores mean higher physical activity level (better outcome).
Time Frame: Baseline and month 18
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the enrolment visit to the last study visit. Since this study terminated early, no adverse event data was to be collected beyond 06 December 2023.
Description: In addition to reporting adverse and serious adverse events, reporting of events of special interest (inhibitor development, thrombotic events,serious hypersensitivity reaction including anaphylactic reactions) was included.
Arm/Group | Efmoroctocog Alfa or Eftrenonacog Alfa
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
Study was terminated early. Only 10 patients had baseline assessments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/66/NCT05856266/Prot_SAP_000.pdf